CLINICAL TRIAL: NCT06722534
Title: Celecoxib for Prevention of Progression in Peutz-Jeghers Syndrome: A Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Celecoxib for Prevention of Progression in Peutz-Jeghers Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY20242368
Record Dates: First submitted 2024-11-12; First posted 2024-12-09 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Peutz-Jeghers Syndrome; Celecoxib; Small Bowel Polyp
MeSH Terms: conditions — Peutz-Jeghers Syndrome | interventions — Celecoxib

STUDY DESIGN:
Intervention Model Description: Participants in the interventional group receive 200 mg celecoxib twice daily for 6 months
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants in the control group receive identically appearing placebo twice daily for 6 months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Celecoxib group (Experimental): Participants in the interventional group receive 200 mg celecoxib twice daily for 6 months
  Interventions: Drug: Celecoxib 400mg
- Placebo group (Active Comparator): Participants in the control group receive identically appearing placebo twice daily for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib 400mg — Participants in the interventional group receive 200 mg celecoxib twice daily for 6 months
  Arms: Celecoxib group
Drug: Placebo — Participants in the control group receive identically appearing placebo twice daily for 6 months
  Arms: Placebo group

SUMMARY:
The Peutz-Jeghers Syndrome (PJS) is a rare autosomal dominant syndrome characterized by mucocutaneous pigmentations, multiple gastrointestinal hamartomatous polyps, and an elevated risk of developing malignancies. Patients with PJS often experience recurrent gastrointestinal polyps that gradually increase in number and size, requiring repeated treatments. As the disease progresses, most patients are forced to undergo multiple surgical or endoscopic treatments. Small bowel polyps develop in 60-90% of patients with PJS, and intussusception occurs in 65% of these patients. Currently, on-demand surgery or scheduled endoscopic polypectomy is the standard of care for the management of small bowel polyps, and among patients who have undergone an initial surgery, reoperation is performed in up to 40% within 5 years. In addition, 8-40% of patients develop small bowel polyp-related complications even with multiple endoscopic treatments. However, surgery and endoscopic treatments are associated with complications, including short bowel syndrome, intestinal adhesions, bowel perforation and bleeding, and health-related quality of life. These problems often lead to decreased patient compliance and even treatment resistance, which increases the risk of disease progression. Because surgical and endoscopic treatment do not completely eliminate the potential for future polyps or extraintestinal neoplasms, there is an unmet medical need for the identification and use of pharmacologic agents to delay endoscopic or surgical interventions.

Cyclooxygenase (COX) is overexpressed in hamartomatous polyp tissue from PJS individuals, which may provide an avenue for possible effective chemoprevention of polyp formation and growth in PJS. Celecoxib, a COX-2 inhibitor, has been shown to reduce polyp burden by 54% in PJS model mice. In addition, the study evaluated the treatment effect of celecoxib on six patients with PJS, two of whom experienced a reduction in gastric polyp burden after six months. These findings provide preliminary evidence that celecoxib may delay the progression of PJS as a potential pharmacological prophylaxis.

Investigators plan to conduct a multicenter, double-blind, randomized, placebo-controlled trial to evaluate the efficacy and safety of celecoxib, and they will use a time-to-event analysis with a composite efficacy end point to determine whether celecoxib can delay disease progression or reduce the need for important endoscopic or surgical procedures in patients with PJS.

ELIGIBILITY:
Inclusion Criteria:

- Patients with PJS ≥ 8 years of age

Diagnostic criteria for PJS: meeting any of the following criteria or presence of an STK11 gene variant:

1. Two or more histologically confirmed PJS hamartomatous polyps;
2. Any number of PJS polyps detected in an individual with a family history of PJS in close relative(s);
3. Characteristic mucocutaneous pigmentation in an individual with a family history of PJS in close relative(s);
4. Any number of PJS polyps in an individual with characteristic mucocutaneous pigmentation.

Exclusion Criteria:

1. Allergy to NSAIDs;
2. Long-term use of any dose of NSAIDs, including aspirin or celecoxib, within 6 months prior to enrollment (willing to undergo a 3-month washout period to restore eligibility);
3. Imaging indicate small intestinal polyps ≥ 3 cm in diameter, intestinal intussusception, intestinal obstruction or intestinal tumor at the time of enrollment;
4. Surgical treatment for small intestinal polyps within 2 years prior to enrollment;
5. Anticipated small bowel resection due to severe polyps within 6 months of enrollment;
6. Receiving other medications for gastrointestinal polyps;
7. Peptic ulcer within 3 months prior to enrollment;
8. Unstable cardiorespiratory condition;
9. Serious renal, hepatic or haematological dysfunction (creatinine >1.5 × ULN; ALT >1.5 × ULN, AST >1.5 × ULN, ALP >1.5 × ULN, TBIL >2 × ULN; haemoglobin <10 g/dL, platelet count <100,000/mL, white blood cells <3000/mL) or other systemic diseases are unsuitable for participation in this study;
10. Pregnancy or breastfeeding;
11. Unwilling or unable to sign the informed consent form

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
The progression of small bowel disease (composite end point) | 2 years
  1. 25% increase in the mean or median diameter of the 5 largest small bowel polyps in abdominal CT/MR (less than 5 polyps will be counted as actual number);
  2. Imaging suggestive small bowel obstruction or small bowel intussusception;
  3. Enteroscopy treatment is required due to the large size of the small bowel polyps or related symptoms;
  4. Surgical treatment is required for intestinal obstruction or intussusception when conservative treatment is ineffective, unresectable small bowel polyps by enteroscopy, or other serious complications associated with small bowel polyps.

SECONDARY OUTCOMES:
Drug-related adverse events (Severity assessed according to CTCAE 5.0) | 2 years
Burden of gastroduodenal and colonic polyps based on gastrointestinal endoscopy (mean or median diameter of 5 largest polyps) | 2 years
Other complications of PJS polyps | 2 years
  1. Gastrointestinal bleeding (hemoglobin drop of 3 g)
  2. Malnutrition (albumin ≤ 35 g/L)
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30（EORTC QLQ-C30） | 2 years
  Changes from baseline by time point in EORTC QLQ-C30 scores
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire ⁃ Colorectal Cancer 29（EORTC QLQ ⁃CR29） | 2 years
  Changes from baseline by time point in EORTC QLQ-CR29 scores
EuroQol Five Dimensions Questionnaire（EQ-5D） | 2 years
  Changes from baseline by time point in EQ-5D scores
Number of enteroscopy or surgical treatments and related complications | 2 years
Incidence of gastrointestinal and other systemic tumors | 2 years
The mortality rate | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Diseases, Air Force Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
Other researchers can contact PI to get IPD.